CLINICAL TRIAL: NCT00015847
Title: A Phase I/II Dose-Finding Study to Determine the Safety, Tolerability, and Anti-Leukemic Effects of STI571 (NSC 716051) in Combination With Interferon-alpha in Patients With Chronic Myelogenous Leukemia in Chronic Phase
Brief Title: Imatinib Mesylate and Interferon Alfa in Treating Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068443; OHSU-6263 (Other: Old OHSU IRB); OHSU-409 (Other: OHSU IRB); NCI-2794; OHSU-HEM-00072-LX
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant interferon alfa — IFN-α will be given at a dose ranging up to 5 MIU daily via subcutaneous injection.
Drug: imatinib mesylate — Once daily oral administration of STI571 (imatinib mesylate) at a dose of 400 mg or 600mg for 12 months.
  Other Names: STI571

SUMMARY:
RATIONALE: Imatinib mesylate and interferon alfa may interfere with the growth of the cancer cells. Combining imatinib mesylate with interferon alfa may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining imatinib mesylate with interferon alfa in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of interferon alfa administered with imatinib mesylate in patients with chronic phase chronic myelogenous leukemia. (Phase I closed to accrual as of 7/9/03.)
* Determine the safety and tolerability of this regimen in this patient population.
* Determine the complete, major, and minor cytogenetic response rates and complete hematologic response rate in patients after 6 and 12 months of treatment with this regimen.
* Determine the molecular response (reverse transcriptase-polymerase chain reaction for bcr-abl) rate in patients who have a complete cytogenetic response after 6 and 12 months of treatment with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

* Phase I (closed to accrual as of 7/9/03): Patients receive oral imatinib mesylate once daily beginning on day 1 and interferon alfa (IFN-A) subcutaneously once daily or 3 times weekly beginning on day 14. Courses repeat every 35 days for up to 1 year in the absence of disease progression or unacceptable toxicity. After completion of 1 year of therapy, patients may receive additional therapy, provided that the patient is benefiting from imatinib mesylate. IFN-A is discontinued in patients who achieve a molecular remission that is confirmed on 2 successive bone marrow samples. Imatinib mesylate is discontinued in patients who achieve and maintain a molecular remission for 2 years.

Sequential dose escalation of IFN-A is followed by sequential dose escalation of imatinib mesylate. Cohorts of 3-6 patients receive escalating doses of IFN-A and then imatinib mesylate until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive imatinib mesylate and IFN-A as in phase I at the established MTD.

Patients are followed for 30 days.

PROJECTED ACCRUAL: Approximately 3-15 patients will be accrued for the phase I portion of this study. (Phase I closed to accrual as of 7/9/03.) A total of 40 patients will be accrued for the phase II portion of the study within 3-4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytogenetically confirmed chronic myelogenous leukemia (CML)

  * Less than 15% blasts in peripheral blood or bone marrow
  * Less than 30% blasts and promyelocytes in peripheral blood or bone marrow
  * Less than 20% basophils in blood or bone marrow
  * Platelet count at least 100,000/mm^3
* No leukemia beyond bone marrow, blood, liver, or spleen
* No chloroma
* Phase I (closed to accrual as of 7/9/03):

  * Philadelphia (Ph) chromosome-positive CML in chronic phase
* Phase II:

  * Newly diagnosed Ph chromosome-positive CML in chronic phase
  * Initial diagnosis within 6 months of study
  * No prior therapy for CML except hydroxyurea and/or anagrelide hydrochloride
* Phase I (closed to accrual as of 7/9/03) and II:

  * No identified sibling donors where allogeneic stem cell transplantation is elected as first-line therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective barrier contraception during and for at least 3 months after study participation
* No other serious uncontrolled medical condition
* No autoimmune disease
* No prior noncompliance to medical regimens or potential unreliability
* No prior grade 3 or greater non-hematologic toxicity due to prior interferon (phase I [closed to accrual as of 7/9/03])

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior bone marrow or peripheral blood stem cell transplantation
* At least 2 weeks since prior interferon alfa (phase I [closed to accrual as of 7/9/03])

Chemotherapy:

* See Disease Characteristics
* At least 6 weeks since prior busulfan (phase I [closed to accrual as of 7/9/03] )
* At least 2 weeks since prior cytarabine (phase I [closed to accrual as of 7/9/03])
* No concurrent chemotherapy
* Concurrent hydroxyurea allowed during the first 3 months of study

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 4 weeks since prior investigational agents other than imatinib mesylate (phase I [closed to accrual as of 7/9/03])
* No concurrent grapefruit juice
* Concurrent anagrelide hydrochloride allowed during the first 3 months of study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Druker, MD, Study Chair — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - OHSU Knight Cancer Institute, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Complete Cytogenetic Response at 6 and 12 Months (Phase II)
Description: Cytogenetic response in terms of the percentage of Ph chromosome positive metaphases in bone marrow is defined as follows:
  Complete* (0% Ph-positive cells) Partial* (1-34%) Minor (35-95%) None (96-100%).
Time Frame: At 6 and 12 months during phase II
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 25
Participants | 13

2. Primary Outcome: Minor Cytogenetic Response at 6 and 12 Months (Phase II)
Time Frame: At 6 and 12 months during phase II
Population: The reason why remaining outcomes can not be reported is due to loss of the study data. Results published 13 years ago were only partial at the time despite having overlapping timeframes with other outcomes. Efforts made since to locate original data to report remaining outcomes were unsuccessful due to early termination and staff turnover.
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

3. Primary Outcome: Complete Hematologic Response at 6 and 12 Months (Phase II)
Time Frame: At 6 and 12 months during phase II
Population: as for outcome 2
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

4. Primary Outcome: Molecular Response in Patients With Complete Cytogenetic Response at 6 and 12 Months (Phase II)
Time Frame: At 6 and 12 months during phase II
Population: as for outcome 2
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 0

5. Primary Outcome: Treatment-related Toxicity (i.e., Grade 3 or 4 Nonhematologic Toxicity) as Measured by NCI CTCAE v3.0 (Phase I)
Description: 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death
Time Frame: 12 Months
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 25
Participants | 8

6. Primary Outcome: Major Cytogenetic Response After 6 and 12 Months of Treatment.
Description: Cytogenetic response in terms of the percentage of Ph chromosome positive metaphases in bone marrow is defined as follows:
  Complete* (0% Ph-positive cells) Partial* (1-34%) Minor (35-95%) None (96-100%).
  *Major cytogenetic response includes complete and partial cytogenetic response.
Time Frame: 6 and 12 months after treatment
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 25
Participants | 18

ADVERSE EVENTS:
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=25)
Fatigue (General disorders) | 1 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (4)
Elevated Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) (Hepatobiliary disorders) | 3 (6)
Infection (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=25)
Chills (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2
Depression (Psychiatric disorders) | 2
Headache (General disorders) | 2
Gout (Musculoskeletal and connective tissue disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination; 12 month follow-up was not carried out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes